CLINICAL TRIAL: NCT01111253
Title: DIABOLO Trial: A Multicenter Randomized Clinical Trial Investigating the Cost-effectiveness of Treatment Strategies With or Without Antibiotics for Uncomplicated Acute Diverticulitis.
Brief Title: Diverticulitis: Antibiotics or Close Observation?
Acronym: DIABOLO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Digestive Diseases Foundation (Other)
Responsible Party: Principal Investigator, M.A. Boermeester, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/233; 2009-015004-26 (EudraCT Number); NL29615.018.09 (Registry Identifier: Nederlands Trial Register (=Dutch Trial Registry)); ABR 29615 (Other: CCMO Registry); 80-82310-97-10039 (Other Grant/Funding Number: ZonMW (Organisation for Health Research and Development)); WO 08-54 (Other Grant/Funding Number: MLDS)
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Diverticulitis
Keywords: multicenter randomized, open label, clinical trial; acute uncomplicated (mild) diverticulitis; treatment strategies; management of diverticulitis; antibiotics; observation and supportive care; cost analysis; economic evaluation
MeSH Terms: conditions — Diverticulitis; Lymphoma, Follicular | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative strategy with antibiotics (Active Comparator): * Hospital admission
  * Intravenous fluids and at least 48 hours of intravenous antibiotics and subsequently switch to oral antibiotics if tolerated (otherwise continuation i.v.) to complete a full 10-day treatment duration
  * Adequate pain relief
  * Oral intake as tolerated
  * Daily monitoring
  Interventions: Drug: Amoxicillin-clavulanate
- Liberal strategy without antibiotics (No Intervention): * Admission only if discharge criteria are not met
  * No initial antibiotics
  * Intravenous fluids only for those not tolerating oral liquids
  * Adequate pain relief
  * Oral intake as tolerated
  * Daily monitoring when admitted to the hospital
  * Self-monitoring at home (Patient diary with temperature and VAS pain score until full recovery)

INTERVENTIONS:
Drug: Amoxicillin-clavulanate — Amoxicillin-clavulanate: 4 times a day 1200 mg and switch to oral administration 3 times a day 625 mg after two days, for a total duration of 10 days.
  In case of allergy to Amoxicillin-clavulanate: intravenous administration ciprofloxacin 2 times a day 400 mg and metronidazole 3 times a day 500 mg. In case of oral administration ciprofloxacin 2 times a day 500 mg and metronidazole 3 times a day 500 mg. For a total duration of 10 days.
  Other Names: Augmentin.
  Arms: Conservative strategy with antibiotics

SUMMARY:
Rationale

The prevalence of colonic diverticular disease is increasing in Western countries. Approximately 10 to 25% of patients with diverticular disease will eventually develop an episode of acute diverticulitis. Currently conservative treatment often includes antibiotic therapy. This advice lacks sound evidence and is merely based on experts' opinion. An old clinical dogma is being clarified with this randomized trial.

Objective

Primary objective is to evaluate whether or not using antibiotics reduces to time to full recovery of an attack of uncomplicated (mild) diverticulitis. Secondary objectives are to evaluate complications, quality of life, readmission rate, recurrence rate, medical and non-medical costs, and antibiotic resistance/sensitivity in both groups.

Hypothesis

The investigators hypothesis is that in the treatment of uncomplicated (mild) acute diverticulitis, supportive treatment without antibiotics is a more cost-effective approach than conservative treatment with antibiotics with respect to time-to-recovery as primary outcome.

Study design

A randomized, open label, multicenter clinical trial comparing treatment of acute uncomplicated diverticulitis with antibiotics to observation and supportive care alone.

Study population

Patients 18 years or older are eligible for inclusion if they have a diagnosis of acute uncomplicated diverticulitis as demonstrated by imaging. Only patients with stages 1a and 1b according to Hinchey's classification or "mild" diverticulitis according to the Ambrosetti criteria are included.

Intervention

Conservative strategy with antibiotics: supportive measures and at least 48 hours of intravenous antibiotics (and therefore admittance to the hospital) and subsequently switch to oral antibiotics if tolerated (total duration of 10 days).

Control

Liberal strategy without antibiotics: supportive measures only. Observation and oral intake as tolerated. Admittance only if discharge criteria are not met on presentation.

Main study parameters/endpoints

The primary endpoint is time-to-recovery with a 6-month follow-up period. Secondary endpoints are occurrence of complicated diverticulitis requiring surgery or percutaneous treatment, morbidity, health related quality of life, readmission rate, recurrence rate, medical and non-medical costs, and antibiotic resistance/sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Only left-sided uncomplicated (mild) acute diverticulitis;
* Clinical suspicion of acute diverticulitis. For acute diagnostic work-up: ultrasound or CT proven diverticulitis. In the case of diverticulitis-negative ultrasound in clinically suspected patients an intravenous contrast-enhanced CT scan is mandatory for confirmation of diverticulitis or exclusion of other pathology. CT for Hinchey/Ambrosetti classification (which is a CT-based classification system) is needed for all patients, but can be delayed 1 day in those with ultrasound diagnosis. Staging diverticulitis is defined according the modified Hinchey/Ambrosetti staging, only stages 1a and 1b and "mild" diverticulitis (1a Confined pericolic inflammation, 1b Confined small (smaller than 5cm) pericolic abscess) are included;
* All patients with informed consent.

Exclusion Criteria:

* Previous radiological (ultrasound and/or CT) proven episode of diverticulitis;
* Colonic cancer;
* Inflammatory bowel disease (ulcerative colitis, Crohn's disease);
* Hinchey stages 2, 3 and 4 or "severe" diverticulitis according to the Ambrosetti criteria, which require surgical or percutaneous treatment;
* Disease with expected survival of less than 6 months;
* Contraindication for the use of the study medication (e.g. patients with advanced renal failure or allergy to antibiotics used in this study);
* Pregnancy, breastfeeding;
* ASA (American Society of Anaesthesiologists) classification > III;
* Immunocompromised patients;
* Clinical suspicion of bacteraemia (i.e. sepsis);
* The inability of reading/understanding and filling in the questionnaires;
* Antibiotic use in the 4 weeks before admittance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 533 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-04 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Time-to-full-recovery | 6 months follow-up

SECONDARY OUTCOMES:
Direct medical costs | 6 months follow-up
Occurrence of complicated diverticulitis defined as abscess, perforation, stricture and/or fistula and need for percutaneous drainage and/or operation | 24 months follow-up
Predefined side-effects of initial antibiotic treatment | 24 months follow-up
  e.g. antibiotic resistance/sensitivity pattern, allergy
Morbidity, like urinary tract infection, pneumonia, etc | 24 months follow-up
Mortality | 24 months follow-up
Readmission rate | 6 months follow-up
Indirect medical costs | 6 months follow-up
Acute diverticulitis recurrence rate | 12 months follow-up
Acute diverticulitis recurrence rate | 24 months follow-up
Health status | 3 months follow-up
  Changes and valuation over time (compared to t=0) will be measured using generic and disease specific quality of life questionnaires (Euro-Qol 5D, Short Form 36 (SF-36) and the Gastro-intestinal Quality of Life Index (Giqli))
Health status | 6 months follow-up
  Changes and valuation over time (compared to t=0 and 3 months) will be measured using generic and disease specific quality of life questionnaires (Euro-Qol 5D, Short Form 36 (SF-36) and the Gastro-intestinal Quality of Life Index (Giqli))
Health status | 12 months follow-up
  Changes and valuation over time (compared to t=0, 3 and 6 months) will be measured using generic and disease specific quality of life questionnaires (Euro-Qol 5D, Short Form 36 (SF-36) and the Gastro-intestinal Quality of Life Index (Giqli))
Health status | 24 months follow-up
  Changes and valuation over time (compared to t=0, 3, 6 and 12 months) will be measured using generic and disease specific quality of life questionnaires (Euro-Qol 5D, Short Form 36 (SF-36) and the Gastro-intestinal Quality of Life Index (Giqli))

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Boermeester, MD, PhD, MSc, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (24):
- Netherlands (24):
  - Ziekenhuisgroep Twente, Almelo
  - Flevo Hospital, Almere Stad
  - Meander Hospital, Amersfoort
  - Academic Medical Center, Amsterdam
  - BovenIJ Hospital, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Sint Lucas Andreas Hospital, Amsterdam
  - Slotervaart Hospital, Amsterdam
  - VU Medical Center, Amsterdam
  - Gelre Hospitals, Apeldoorn
  - Rijnstate Hospital, Arnhem
  - Rode Kruis Hospital, Beverwijk
  - Reinier de Graaf Gasthuis, Delft
  - Albert Schweitzer Hospital, Dordrecht
  - Kennemer Hospital, Haarlem
  - Ziekenhuisgroep Twente, Hengelo
  - Tergooi Hospital, Hilversum
  - Spaarne Hospitals, Hoofddorp
  - Westfries Gasthuis, Hoorn
  - Sint Antonius Hospital, Nieuwegein
  - Erasmus Medical Center, Rotterdam
  - Ikazia Hospital, Rotterdam
  - Sint Franciscus Gasthuis, Rotterdam
  - Máxima Hospital, Veldhoven

REFERENCES:
- [Background] de Korte N, Unlu C, Boermeester MA, Cuesta MA, Vrouenreats BC, Stockmann HB. Use of antibiotics in uncomplicated diverticulitis. Br J Surg. 2011 Jun;98(6):761-7. doi: 10.1002/bjs.7376. Epub 2011 Jan 6. PMID 21523694
- [Background] de Korte N, Kuyvenhoven JP, van der Peet DL, Felt-Bersma RJ, Cuesta MA, Stockmann HB. Mild colonic diverticulitis can be treated without antibiotics. A case-control study. Colorectal Dis. 2012 Mar;14(3):325-30. doi: 10.1111/j.1463-1318.2011.02609.x. PMID 21689302
- [Background] de Korte N, Klarenbeek BR, Kuyvenhoven JP, Roumen RM, Cuesta MA, Stockmann HB. Management of diverticulitis: results of a survey among gastroenterologists and surgeons. Colorectal Dis. 2011 Dec;13(12):e411-7. doi: 10.1111/j.1463-1318.2011.02744.x. PMID 21819518
- [Background] Unlu C, de Korte N, Daniels L, Consten EC, Cuesta MA, Gerhards MF, van Geloven AA, van der Zaag ES, van der Hoeven JA, Klicks R, Cense HA, Roumen RM, Eijsbouts QA, Lange JF, Fockens P, de Borgie CA, Bemelman WA, Reitsma JB, Stockmann HB, Vrouenraets BC, Boermeester MA; Dutch Diverticular Disease 3D Collaborative Study Group. A multicenter randomized clinical trial investigating the cost-effectiveness of treatment strategies with or without antibiotics for uncomplicated acute diverticulitis (DIABOLO trial). BMC Surg. 2010 Jul 20;10:23. doi: 10.1186/1471-2482-10-23. PMID 20646266
- [Background] Draaisma WA, van de Wall BJ, Vermeulen J, Unlu C, de Korte N, Swank HA. [Treatment for diverticulitis not thoroughly researched]. Ned Tijdschr Geneeskd. 2009;153:A648. Dutch. PMID 19857313
- [Background] Unlu C, Daniels L, Vrouenraets BC, Boermeester MA. A systematic review of high-fibre dietary therapy in diverticular disease. Int J Colorectal Dis. 2012 Apr;27(4):419-27. doi: 10.1007/s00384-011-1308-3. Epub 2011 Sep 16. PMID 21922199
- [Derived] Daniels L, Unlu C, de Korte N, van Dieren S, Stockmann HB, Vrouenraets BC, Consten EC, van der Hoeven JA, Eijsbouts QA, Faneyte IF, Bemelman WA, Dijkgraaf MG, Boermeester MA; Dutch Diverticular Disease (3D) Collaborative Study Group. Randomized clinical trial of observational versus antibiotic treatment for a first episode of CT-proven uncomplicated acute diverticulitis. Br J Surg. 2017 Jan;104(1):52-61. doi: 10.1002/bjs.10309. Epub 2016 Sep 30. PMID 27686365